CLINICAL TRIAL: NCT03932825
Title: A Clinical Trial of Nitrous Oxide for Treatment-Resistant Major Depressive Disorder
Brief Title: Nitrous Oxide for Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lingjiang Li (Other)
Responsible Party: Sponsor-Investigator, Lingjiang Li, President of Chinese Psychiatry Society of Chinese Medical Association, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-05-04-XY-0001
Record Dates: First submitted 2019-04-20; First posted 2019-05-01 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Depressive Disorder; Major Depressive Disorder; Treatment Resistant Depression; Depressive Disorder, Major; Depression
Keywords: Nitrous Oxide; Laughing Gas
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — Nitrous Oxide; xiao-cheng-qi-tang

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Air oxygen mixture (Placebo Comparator): participants in this arm inhale mixed oxygen-air gas (inspired oxygen concentration ~50%).
  Interventions: Drug: Placebo
- Nitrous oxide (Experimental): Participants in this group inhale mixed 50% nitrous oxide and 50% oxygen.
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — An 1-hour session of inhaled nitrous oxide at concentrations of 50%.
  Other Names: Laughing Gas; Xiao Qi; 笑气
  Arms: Nitrous oxide
Drug: Placebo — An 1-hour session of mixed oxygen-air gas(inspired oxygen concentration ~50%)
  Other Names: Air oxygen mixture
  Arms: Air oxygen mixture

SUMMARY:
This study aims at investigating the persistence of antidepressant effect of Nitrous Oxide (N2O) for Treatment-Resistant Depression(TRD). The investigators also aim to assess the effect of N2O on the electroencephalograph, multimodal magnetic resonance imaging(MRI), blood cytokines, feces bacteria flora and neuropsychological performance in patients with TRD. The investigators further aim to identify the predictors of N2O's antidepressant effeect using the above techniques.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years, both sexes), with ICD-10 criteria for MDD without psychosis, as determined by a structured clinical interview Mini International Neuropsychiatric Interview
* Moderate to severe depression, as defined by a pretreatment score >17 on the HDRS-17 scale
* TRD was defined as having had at least two adequate dose-duration, antidepressant medication failures in the current episode and a lifetime failure of at least three antidepressant medication trials.
* Informed consent to participate in this study

Exclusion Criteria:

* A history of bipolar disorder, schizophrenia, schizoaffective disorder, obsessive-compulsive disorder, panic disorder, or documented Axis II diagnoses; active suicidal intention, as determined by clinical interview
* Active or recent (<12 months) substance abuse or dependence; excluding nicotine
* Presence of acute medical illness that could interfere with study participation, including significant pulmonary disease
* Acute severe suicidal ideation
* Acute psychosis
* Received ECT treatment within 6 months
* History of NMDA-antagonists (e.g., ketamine) intake
* Pregnancy or breastfeeding
* Any contraindications to the use of nitrous oxide (e.g., pneumothorax, middle ear occlusion, elevated intracranial pressure, chronic cobalamin or folate deficiency unless treated with folic acid or vitamin B12).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale-17 item (HDRS-17) | Baseline, 2hours, 24hours, 7days, 2weeks
  Interview-based questionnaire used to measure the severity of depression. Consists of 17 items with a score calculated. Higher scores are associated with more severe depression.
  0 - 7 = Normal; 8 - 17 = Mild Depression; 18 - 24 = Moderate Depression; > 25 = Severe Depression; Maximum score = 52
Change in QIDS-16-SR (Quick Inventory of Depressive Symptomatology-16 Self Report) | Baseline, 2hours, 24hours, 7days, 2weeks
  This is a 16-item self report questionnaire that measures depressive symptoms. Improvement is reported in change in depressive score score ranges from 0-27, with higher numbers indicating more severe symptom reporting.
  Change is calculated by baseline plus/minus the value at the later time point
Change in Visual Analog Scale-Depression (VAS-D) | Baseline, 2hours, 24hours, 7days, 2weeks
  All patients are asked to fill out visual analog scale for depression (VAS-D) before and after the intervention. VAS-D is a self-report scale for ddepression severity, with 0 score indicating not at all depressed and 10 score indicating extremely depressed.

SECONDARY OUTCOMES:
Chang in Event Related Potentials (ERPs) | Baseline, 24hours, 7days, 2weeks
  The investigator employ 64-lead Event Related Potentials (ERPs) to assess the resting-state EEG signal and signals during specific neurocognitive processes related to tasks, including an emotional face recognition task, a dot probe task and a self-referential personality word memory task.
Change in voxel-based morphometry of grey matter, white matter as assessed by structural magnetic resonancce imaging. | Baseline, 24hours
  Participants will receive resting-state functional magnetic resonance imaging (MRI). Scans will be performed on a 3.0-T Siemens Magnetom Skyra scanner (Siemens Healthineers, Erlangen, Germany). During scanning, all participants were instructed to remain motionless, and to think of nothing in particular but to not fall asleep.
Change in Functional connectivity | Baseline, 24hours
  Change in Functional connectivity of the brain networks between baseline and after the inhaled Nitrous oxide 24hours as assessed by measure of connectivity in multimodal MRI.
Change in peripheral blood cytokines | Baseline, 2hours, 24hours
  Peripheral blood sample will be collected and the concentration of IL-6, TNF-α, and CRP will be assessed.
Change in feces bacterial flora | Baseline
  The objective of investigator is to characterize gut microbiome in patients with TRD. To explore the specific diversity of gut microbiome.
  The stool samples were collected in the collection kits at the baseline, and were frozen at -80 °C. After the process of DNA Purification, 16S rRNA Gene Amplification and Illumina MiSeq sequencing, the study finally find the abundance and diversity of microbiota.
Change in the TMT/A and B (Executive Function) | Baseline, 24hours, 7days, 2weeks
  Trail Making Test (TMT) is a cognitive test designed to assess scanning, visuomotor tracking, executive function, and cognitive flexibility. It consists of two parts, A and B: the patient must draw lines to connect consecutively numbered circles (part A) and then connect consecutively numbered and lettered circles alternating between the two sequences (part B). The time taken to complete the two parts is recorded. Part A assesses cognitive processing speed. The lower the score the faster the processing speed.
Change in Congruent STROOP Time to Complete (Executive Function) | Baseline, 24hours, 7days, 2weeks
  Stroop Colour Naming Test (STROOP) is a cognitive test designed to assess the ability to inhibit a prepotent response to reading words while performing a task that requires attention control. It comprises two sheets with 50 words on each, and each word is the name of a colour. On the first sheet, the Congruent STROOP Sheet, the word and ink colour match; on the Incongruent STROOP Sheet, the word and ink colour do not match. For each sheet, the patient has 4 minutes to name the ink colour of each word. When the patient finishes the sheet, or once 4 minutes is up, the clinician notes the time taken and counts the number of correct and incorrect responses. The scale ranges from 0-100, the higher score the greater the cognitive flexibility.
Digit-Span Test | Baseline, 24hours, 7days, 2weeks
  Score range 0-12 for each of for dimensions: Digit span forward, digit span backward, block span forward, block span backward. Higher scores indicate better cognitive performance.
Change in DSST (Number of Correct Symbols) | Baseline, 24hours, 7days, 2weeks
  Digit Symbol Substitution Test (DSST) is a cognitive test designed to assess psychomotor speed of performance requiring visual perception, spatial decision-making, and motor skills. It consists of 133 digits and requires the patient to substitute each digit with a simple symbol in a 90-second period. Each correct symbol is counted, and the total score ranges from 0 (less than normal functioning) to 133 (greater than normal functioning)." as a description of DSST.
Improvement on Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline, 2hours, 24hours, 7days, 2weeks
  The Snaith-Hamilton Pleasure Scale (SHAPS) assesses the anhedonia symptoms of MDD patients, with higher score indicating more severe anhedonia.
  Evaluating the patient's pleasure experience and choosing the degree of agreement with the happy response in some pleasant situations, and each item was rated on a 4-point scale."1 = Strongly agree, 2 = agree, 3 = disagree and 4 = strongly disagree" This scale evaluates the status of patients in the recent period of time, The total score of the scale is the sum of the scores of 14 items, with a total score of 14-56. The higher the total score, the more serious the anhedonia.
Change in Hamilton Anxiety Rating Scale (HAM-A) | Baseline, 2hours, 24hours, 7days, 2weeks
  Assessed via the Hamilton Anxiety Rating Scale (HAM-A). The HAM-A score ranges from 0 (no present anxiety) to 56 (maximum anxiety score).

OTHER OUTCOMES:
Change in Heart Rate Variability | Baseline, 2hours, 24hours, 7days, 2weeks
  The investigator will assess the heart rate variability (HRV) of all participants before and after the intervention.
Number of Participants With Adverse Events AEs | Baseline, 2hours, 24hours, 7days, 2weeks
  AEs are any untoward, undesired, or unplanned event in the form of signs, symptoms, disease, or laboratory or physiologic observations occurring in a person given study treatment. The event does not need to be causally related to the study treatment.
Clinician-Administered Dissociative States Scale (CADSS) Scores During inhaled nitrous oxide | Baseline, 2hours, 24hours
  The CADSS is a 23-item self-report scale for the assessment of dissociative states. It is a reliable, valid self-report instrument. The severity of each dissociative symptom ranges from 0 (not present) to 4 (extreme). The total score is calculated by summing across items, with a total possible range of 0-92. The CADSS was administered right before inhaled, and 2hours and 24hours after the inhaled. The timeframe is "at this moment".
  Change From Baseline in Clinician-Administered Dissociative States Scale (CADSS) Score.
Suicidal ideation as assessed by the Scale for Suicide Ideation (SSI) | Baseline, 2hours, 24hours, 7days, 2weeks
  The scale contains 19 items rated on a scale from 0 to 2, allowing score range from 0 to 38, score over 4 (first five items) will be considered inclusion criteria. Higher values indicate worsening or presence of suicidal ideation.
  Item 4 and 5 at the end of the last week was assessed. If the answer to both questions was "no", the patient was judged to have no suicidal ideation.If either answer is "weak" or "moderate to strong," it is considered suicidal ideation.The intensity of suicidal ideation was judged according to the mean value of items 1-5 in the scale. The higher the score, the greater the intensity of suicidal ideation.The risk of suicide was assessed according to items 6-19 of the suicide ideation scale.The total score was calculated by [(the sum of item 6-19 scores -9)/33]*100. The higher the score, the greater the risk of suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Lingjiang Li, MD, Principal Investigator — Mental Health Institute, the Second Xiangya Hospital of Central South University
Locations (1):
- Mental Health Institute & Faculty of Psychiatry of The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No